CLINICAL TRIAL: NCT05304234
Title: Liver Cancer Disparities in American Indian and Alaska Native Persons
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Cherokee Nation Health Services (Unknown); Alaska Native Tribal Health Consortium (Other)
Responsible Party: Principal Investigator, George Ioannou, Professor, School of Medicine, Gastroenterology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STUDY00013583; 1P20CA252732-01A1 (NIH)
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Hepatocellular Carcinoma; Cirrhosis, Liver; Hepatitis B
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis; Hepatitis B | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: we are performing a pilot and feasibility randomized controlled trial (RCT) of HCC screening by US + AFP every 6 months (n=100), the current standard-of-care, versus aMRI + AFP every 6 months (n=100) for 12 months (i.e. at time 0, 6 and 12 months) among AI/AN patients with cirrhosis or HBV.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound + AFP (Active Comparator): Screening by abdominal ultrasound + serum AFP testing at 0, 6 and 12 months
  Interventions: Diagnostic Test: Ultrasound or abbreviated MRI
- aMRI + AFP (Active Comparator): Screening by abbreviated MRI of the abdomen + serum AFP testing at 0, 6 and 12 months
  Interventions: Diagnostic Test: Ultrasound or abbreviated MRI

INTERVENTIONS:
Diagnostic Test: Ultrasound or abbreviated MRI — Abdominal ultrasound or abbreviated MRI

SUMMARY:
We are performing a pilot and feasibility randomized controlled trial (RCT) of HCC screening by US + AFP every 6 months (n=100), the current standard-of-care, versus aMRI + AFP every 6 months (n=100) for 12 months (i.e. at time 0, 6 and 12 months) among AI/AN patients with cirrhosis or HBV.

DETAILED DESCRIPTION:
We are performing a pilot and feasibility randomized controlled trial (RCT) of HCC screening by US + AFP every 6 months (n=100), the current standard-of-care, versus aMRI + AFP every 6 months (n=100) for 12 months (i.e. at time 0, 6 and 12 months) among AI/AN patients with cirrhosis or HBV.

We will compare the aMRI vs. the US arm with respect to the following outcomes:

1. Compliance/feasibility of conducting all three screening tests (0, 6 and 12 months) - Primary Outcome
2. Proportion of screening tests conducted that employed the appropriate screening protocol and used appropriate documentation of findings with the LI-RADS system - Primary Outcome
3. Proportion diagnosed with HCC and stage at diagnosis - Secondary Outcome

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis, any etiology, or chronic HBV infection
* High risk of HCC
* Age 18-75
* Competent to provide informed consent

Exclusion Criteria:

* Prior diagnosis of HCC
* Current suspicion of HCC
* Prior receipt of any organ transplantation
* Participation in another HCC screening trial
* CTP score >=10
* MELD-Na score >20
* GFR<30
* Poor life expectancy (<5 years)
* Contraindication to MRI
* Inability to complete study visits
* Currently pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Compliance with screening protocol | 12 months
  Compliance with conducting all three screening tests
Feasibility of screening protocol | 12 months
  Proportion of screening tests conducted that employed the appropriate screening protocol and used appropriate documentation of findings with the LI-RADS system

CONTACTS AND LOCATIONS:
Overall Officials: George Ioannou, MD, MS, Principal Investigator — University of Washington
Locations (1):
- Cherokee Nation Health Service, Tahlequah, Oklahoma, United States